CLINICAL TRIAL: NCT04518826
Title: A Comparison Between Fractional Flow Reserve Guided and Coronary Angiography Guided Treatment Using Drug Eluting Balloon in In-stent Restenosis of Drug Eluting Stent: a Single-center, Prospective, Randomized Controlled Clinical Trial
Brief Title: A Comparison Between FFR Guided and CAG Guided Treatment Using DEB in ISR of DES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FFRCAG
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: In Stent Restenosis; Drug Eluting Stent; Coronary Artery Disease
Keywords: fractional flow reserve; in stent restenosis; drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FFR: In FFR group, FFR at maximum hyperemia will be measured after pretreatment of DES-ISR lesion by balloons(non-compliant balloon, cutting balloon or scoring balloon). If FFR <0.9, the operator will dilate the DES-ISR lesion again before another FFR is measured. If FFR>=0.9, DEB will be used and final FFR will be measured at the end of the procedure.
  Interventions: Device: fractional flow reserve
- CAG: In angiography group, the operator will treat the DES-ISR lesion with balloons(non-compliant balloon, cutting balloon or scoring balloon), and then DEB without FFR guidance.

INTERVENTIONS:
Device: fractional flow reserve — FFR is a physiological functional parameter indicating the severity of ischemic myocardium perfused by a diseased coronary artery. It is measured by a pressure wire placed in the coronary artery and calculated by the ratio of pressures distal and proximal to the stenosis.
  Groups: FFR

SUMMARY:
This is a prospective single center, randomized controlled clinical study aimed to compare the clinical and angiographic follow-up results of patients with in-stent restenosis(ISR) after coronary drug eluting stent(DES) implantation treated by fractional flow reserve -guided and angiography guided drug eluting balloon(DEB) intervention. This study intends to confirm the clinical benefits of optimizing DEB intervention of DES-ISR by FFR.

DETAILED DESCRIPTION:
420 patients with DES-ISR will be recruited in this study. After angiography, patients with DES-ISR to be treated with DEB will be randomly assigned to FFR-guided and angiography-guided groups. In FFR group, FFR at maximum hyperemia will be measured after pretreatment of DES-ISR lesion by balloons(non-compliant balloon, cutting balloon or scoring balloon). If FFR <0.9, the operator will dilate the DES-ISR lesion again before another FFR is measured. If FFR>=0.9, DEB will be used and final FFR will be measured at the end of the procedure. In angiography group, the operator will treat the DES-ISR lesion with balloons(non-compliant balloon, cutting balloon or scoring balloon), and then DEB without FFR guidance.

ELIGIBILITY:
Inclusion Criteria:

In-stent restenosis(ISR) occurred more than 6 months after drug eluting stent (DES) implantation

Exclusion Criteria:

1. ISR in bare metal stents and biodegradable stents
2. Complicated with immune diseases
3. ISR in left main DES
4. Suffer from renal failure requiring dialysis treatment or is undergoing dialysis treatment
5. Severe cardiac insufficiency (LVEF <30%)
6. Subjects with ST segment elevation myocardial infarction within 7 days of onset of chest pain
7. Pregnant or lactating women
8. Combined with other diseases, life expectancy <1 year
9. Follow - up visits required by the protocol cannot be followed, or the investigators believe that the participation of subjects in the trial will increase the risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease and DES implantation.
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
target vessel failure | 12 month
  cardiac death, target vessel myocardial infarction, target vessel failure

SECONDARY OUTCOMES:
angiographic outcomes | 12 month
  diameter stenosis, binary stenosis and late lumen loss measured by QCA
target vessel failure | 36 month
  cardiac death, target vessel myocardial infarction, target vessel failure

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No